

#### **ACCUMULATE STUDY**

ImpACt of very high protein Content enteral nUtrition formulas on protein metabolism and residual gastric volume in critically ill MUltipLe trAuma paTiEnts

# - ACCUMULATE trial -

NCT: 05647135

December 1, 2022

# ROSPĖŅ.

#### **ACCUMULATE STUDY**

## Sample size calculation:

- Expected difference ( $\Delta\Delta$ ) = 0.4 g/kg BW
- Standard deviation ( $\sigma\sigma$ ) = 0.5 g/kg BW
- Significance level ( $\alpha \alpha$ ) = 0.05
- Power  $(1-\beta 1-\beta) = 0.80$
- With an expected difference of 0.4 g/kg BW and a standard deviation of 0.5, a minimum sample size of 25 per group is required.
- To ensure robustness and account for drop-outs and variability, targeting at least 28 participants per group is recommended.

### **Statistical Analysis:**

#### 1. Descriptive Statistics:

Summary statistics (mean, standard deviation, median, interquartile range)
will be provided for all continuous variables. Frequencies and percentages will be provided for categorical variables.

#### 2. Primary Outcome Analysis:

- Differences in protein and calorie intake between the groups at day 5 and day 10 will be analyzed using independent t-tests or Mann-Whitney U tests, depending on the data distribution.
- o Differences in residual gastric volume between the groups at day 5 and day 10 will be analyzed using independent t-tests or Mann-Whitney U tests.

#### 3. Secondary Outcome Analysis:

- o Changes in quadriceps rectus femoris thickness over time will be analyzed using repeated measures ANOVA or mixed-effects models.
- Differences in body composition parameters (Fat-Free Mass, Total Body Water, Phase Angle) will be analyzed using paired t-tests or Wilcoxon signedrank tests for within-group comparisons and independent t-tests or Mann-Whitney U tests for between-group comparisons.
- Differences in plasmatic levels of prealbumin and C-reactive protein will be analyzed using independent t-tests or Mann-Whitney U tests.
- Differences in handgrip strength will be analyzed using paired t-tests or Wilcoxon signed-rank tests for within-group comparisons and independent ttests or Mann-Whitney U tests for between-group comparisons.

#### 4. Missing Data:

Missing data will be handled using multiple imputation or other appropriate methods. Sensitivity analyses will be conducted to assess the robustness of the results.

#### 5. Statistical Software:

 All analyses will be performed using statistical software such as SPSS, GraphPad